CLINICAL TRIAL: NCT01319240
Title: A Trial to Investigate Pharmacokinetics, Safety and Tolerability of Insulin Degludec/Liraglutide (A3) Compared With Insulin Degludec and Liraglutide in Healthy Subjects
Brief Title: Safety and Tolerability of Insulin Degludec/Liraglutide (A3) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-3871; 2010-021190-36 (EudraCT Number); U1111-1119-2417 (Other: WHO)
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec; IDegLira; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDegLira (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- IDeg (Active Comparator)
  Interventions: Drug: insulin degludec
- Lira (Active Comparator)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec — Subjects will be randomised to one out of six possible treatment sequences. Single dose, administered subcutaneously (under the skin) on three separate dosing visits.
  Arms: IDeg
Drug: insulin degludec/liraglutide — Subjects will be randomised to one out of six possible treatment sequences. Single dose, administered subcutaneously (under the skin) on three separate dosing visits.
  Arms: IDegLira
Drug: liraglutide — Subjects will be randomised to one out of six possible treatment sequences. Single dose, administered subcutaneously (under the skin) on three separate dosing visits.
  Arms: Lira

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the bioavailability of insulin degludec and liraglutide, when administered either combined or as separate administrations.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Body Mass Index (BMI) between 20.0 and 27.0 kg/m^2 (both inclusive)
* Body weight between 75 kg and 90 kg (both inclusive)
* Fasting plasma glucose below 6.1 mmol/L (110 mg/dL)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as randomised
* Previous participation in any other clinical trial involving other investigational products within the last 3 months before dosing in this trial
* Donation of any blood or plasma in the past month or in excess of 500 mL within the 3 month preceding screening (trial start) or surgery or trauma with more than 500 mL blood loss within the 3 month preceding screening
* History of or presence of cancer, or any clinically significant cardiovascular, respiratory,metabolic, renal, hepatic, gastrointestinal, endocrine, diabetes, haematological, dermatological,venereal, neurological, psychiatric diseases or other major disorders that might have impact on the trial, as judged by the Investigator (Trial Physician)
* Clinically significant abnormal haematology, biochemistry, lipids, urinalysis or coagulation screening tests, as judged by the Investigator (Trial Physician)
* Known hepatitis or known carrier of the hepatitis B surface antigen (HBsAg) or hepatitis C antibodies, or a positive result to the test for HIV (human immunodeficiency virus) antibodies and antigen
* Family or personal history of MEN2 (Multiple endocrine neoplasia syndrome type 2) or familial medullary thyroid carcinoma (FMTC)
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Supine blood pressure at screening, after resting for 5 min, outside the range of 90-140 mmHg systolic or 50-90 mmHg diastolic (excluding white-coat hypertension; therefore, if a repeated measurement on a second screening visit shows values within the range, the subject can be included in the trial) or resting heart rate outside the range of 40-90 bpm
* Clinically significant abnormal ECG (Electrocardiogram) at screening (trial start)
* Significant history of alcoholism or drug/chemical abuse, or a positive result of the urine drug screen or alcohol breath test, or consuming more than 21 units of alcohol per week (one unit of alcohol equals about 250 mL of beer or lager, one glass of wine, or 20 mL spirits)
* Smoking more than 5 cigarettes, or the equivalent, per day and unable to refrain from smoking during the in-house periods
* Mental incapacity or language barriers which preclude adequate understanding or cooperation,unwillingness to participate in the trial or subjects that in the opinion of Investigator (trial physician) should not participate in the trial
* Use of any prescription or non-prescription medication, except for paracetamol, acetylsalicylic acid, and vitamins (but including mega-dose vitamin therapy, as judged by the Investigator (trial physician)) within 2 weeks before the trial
* Any condition that would interfere with trial participation or evaluation of results, as judged by the Investigator (trial physician)
* Subjects with a history of deep leg vein thrombosis or with frequent appearance of deep leg vein thrombosis in 1st degree relatives as judged by the Investigator (trial physician)
* Males who are sexually active and not surgically sterilised, who or whose partner are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Baseline (screening) calcitonin level above or equal to 50 ng/L
* Suffer from a life threatening disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The area under insulin degludec concentration-time curve | from 0-infinity hours after trial product administration
The area under liraglutide concentration-time curve | from 0-infinity hours after trial product administration

SECONDARY OUTCOMES:
The area under insulin degludec concentration-time curve | from 0-120 hours after trial product administration
The area under liraglutide concentration-time curve | from 0-72 hours after trial product administration
Maximum concentration of insulin degludec | from 0-120 hours after trial product administration
Maximum concentration of liraglutide | from 0-72 hours after trial product administration
Number of hypoglycaemic episodes | From day 0 to 7-14 days after 3rd trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com